CLINICAL TRIAL: NCT04134598
Title: ExclUsive endocRine Therapy Or Radiation theraPy for Women Aged ≥70 Years With Luminal A-like Early Stage Breast Cancer (EUROPA): a Randomized Phase 3 Trial
Brief Title: ExclUsive endocRine Therapy Or Radiation theraPy for Women Aged ≥70 Years Early Stage Breast Cancer
Acronym: EUROPA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Icro Meattini, MD, M.D., Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUROPA
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Partial Breast Irradiation; Radiation Therapy; Endocrine Therapy; Breast Conserving Surgery; Elderly; Health Related Quality of Life; Patients Reported Outcome Measures; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Tamoxifen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breast Irradiation (RT) (Experimental): Breast Irradiation (RT)
  Interventions: Radiation: Breast irradiation (RT)
- Endocrine Therapy (ET) (Active Comparator): Endocrine Therapy (ET)
  Interventions: Drug: Endocrine Therapy (ET): letrozole, anastrozole, exemestane, tamoxifen

INTERVENTIONS:
Radiation: Breast irradiation (RT) — Irradiation of volume's portion Index quadrant) or whole volume of the residual breast.
  Other Names: Partial Breast Irradiation (PBI); Whole Breast Irradiation (WBI)
  Arms: Breast Irradiation (RT)
Drug: Endocrine Therapy (ET): letrozole, anastrozole, exemestane, tamoxifen — Adjuvant endocrine therapy as per local policy (letrozole/anastrozole/exemestane/tamoxifene for 5-year or switch schedules aromatase inhibitors/tamoxifen for 5-year).
  Other Names: Hormonal therapy
  Arms: Endocrine Therapy (ET)

SUMMARY:
Rationale and relevance for patients and the scientific community. In low risk early stage patients ≥70 years, exclusive radiation therapy (RT) approach might be superior in terms of Health-Related Quality of Life (HRQoL), when compared to exclusive endocrine therapy (ET) following breast-conserving surgery (BCS). Assuming an equal rate of disease control, unnecessary long-term toxicity of ET may be avoided.

DETAILED DESCRIPTION:
Study Background. BCS has been established as the preferred treatment option for early stage breast cancer (BC) or for initially inoperable tumors that respond sufficiently to preoperative therapy. BCS plus RT obtains at least the same results in terms of survival, without the huge impact on the patient's body image and HRQoL as that seen after mastectomy. For decades, standard whole breast irradiation (WBI) consisted of 45-50 Gy delivered at 1.8-2.0 Gy/fraction over 4.5-5 weeks with or without a boost dose to the surgical bed. Large phase 3 trials evaluating different hypofractionation schedules proved that overall treatment time could be reduced without compromising local control and safety profile.In April 2020, the results of the FAST-Forward phase 3 trial demonstrated the efficacy and safety of a further reduction in the number of treatment fractions to five in one week (26 Gy in 5 fractions) as WBI treatment.

Following the 2022 European Society for Radiotherapy and Oncology Advisory Committee in Radiation Oncology Practice (ESTRO- ACROP) consensus recommendations on patient selection and dose and fractionation for external beam RT in early BC, (1) moderate hypofractionated WBI should be offered regardless of extent of target volumes, age at BC diagnosis, pathological tumor stage, BC biology, surgical margins status, tumor bed boost, breast size, invasive or pre-invasive ductal carcinoma in situ (DCIS) disease, oncoplastic BCS, and use of systemic therapy, and (2) ultra-hypofractionated (26 Gy in five fractions) WBI can be offered as standard of care or within a randomized controlled trial or prospective registration cohort for WBI and for chest wall RT.

Partial breast irradiation (PBI) has been introduced as an alternative treatment method for selected patients with early stage BC. Potential advantages of accelerated PBI include shorter treatment time, equivalent disease control, improved safety profile, and cost reduction as compared to standard WBI. The role of PBI has been investigated in large-scale prospective phase 3 clinical trials (i.e., NSABP-B29/RTOG 0413, IRMA, RAPID, IMPORT-LOW, GEC-ESTRO trials).

5-year results of the IMPORT-LOW trial showed non-inferiority of PBI when compared to WBI in women with low risk early BC, with a 5-year local recurrence (LR) rate of 0.5%. Ongoing research explores other modalities of RT that will minimize toxicities without reducing effectiveness. Intensity-modulated radiotherapy (IMRT) has the theoretical advantage of a further increase in dose conformity compared with three-dimensional techniques, with increased normal tissue sparing. To date, only the Florence IMRT-APBI phase 3 trial reported the outcomes of exclusive IMRT accelerated PBI compared to WBI, demonstrating no significant difference between the two groups in terms of ipsilateral breast tumor recurrences (IBTR). The PBI group presented significantly better results considering acute (p=0.0001), late (p=0.004), and cosmetic outcome (p=0.045). The subgroup analysis evaluating patients aged 70 years or older, showed a 5-year IBTR rate of 1.9% for both groups, and significantly better results in terms of acute skin toxicity, in favor of the PBI arm. Therefore, a significant impact on patients' compliance to RT could translate into a consistent improvement of overall HRQoL.

Heart exposure to ionizing radiation during RT for BC increases subsequent rates of ischemic heart disease (IHD). The increase is proportional to the mean dose to the heart. Women with pre-existing cardiac risk factors have greater absolute increases in risk from RT. An age >70 years seems to be one of the most significant factor for IHD occurrence. PBI represents one of several effective strategies to reduce cardiac radiation dose when compared to WBI.

Postoperative RT in the elderly is a matter of constant debate. RT was shown to benefit these patients with regards to local control; however, the absolute benefit is small (for low risk subtypes). Moreover, considering the poor compliance of elderly patients to conventional RT treatment time (3-6 weeks), conventional RT is often omitted in cases of low-risk BC, at the expense of reducing the local control rate by less than 4%.

In an unplanned subgroup analysis of the PRIME-II trial by estrogen receptor (ER) score, LR at 5 years for women in the rich ER subgroup was lower than in the whole population; for patients assigned no RT, 3% had a LR compared with 1% of women allocated WBI (5-year IBTR was 3.3%, and 1.2%, respectively).

The British Association of Surgical Oncology (BASO)-II trial confirmed that patients treated with either exclusive adjuvant RT or ET with tamoxifen had an equivalent LR rate per year of 0.8%. These data suggested that RT or ET alone resulted in excellent disease control in older women with early BC, and that the combination of treatments may have less benefit than expected. A direct comparison between PBI or ET omission as adjuvant treatment is lacking in the existing literature.

Conversely, the toxicity profile of ET is well known, and could significantly impact long term HRQoL of these potentially frail patients. Elderly patients with early BC are a unique population with regards to good prognosis and potential comorbidities, thus minimizing treatment to maintain HRQoL without compromising survival is extremely important. In the decision-making process for adjuvant therapy, estimates of the patient's risk of benefit and/or harm with treatment should be performed together with an assessment of baseline comorbidities, life expectancy and care preferences. Many large phase III studies reported on the detrimental effects of postmenopausal ET on bone density and fractures incidence, thromboembolic complications, sexual, and cognitive functionality. Moreover, patient's compliance and oral treatment adherence may be a concern, and some patients would like to avoid the toxicities associated with ET.

Considering that the potential benefit of PBI alone could be better than that of the RT-only effect reported in the above WBI-using trials, it may be possible to avoid the long term toxicity of ET and favorably impact HRQoL in selected patients, such as elderly patients with a good prognosis.

Importantly, all previously published de-escalation studies were designed and performed in order to evaluate RT omission, regardless of efficacy and compliance of ET. When expecting a comparable efficacy among tested treatment modalities, HRQoL might be the factor with the most influence on the treatment decision-making process and should therefore be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥70 years;
* histologically proven invasive adenocarcinoma of the breast;
* pathological T1 (pT1) stage (clinical T1-2 [cT1-2] stage is allowed);
* clinical and pathological N0 (cN0 and pN0) stage (isolated tumor cells [i+] allowed);
* any tumor grade (if pT ≤10 mm), G1-2 tumor grade (if pT between 11 and 19 mm);
* Luminal-A by immunohistochemistry (IHC)-based on local assessment (consistent with 14th St. Gallen consensus definition):

  * ER/PgR+ (defined as ≥10% by IHC staining),
  * Human epidermal growth factor receptor 2 (HER2)- (0 or 1+ following IHC staining and proven negative by in-situ hybridization [ISH] in case of 2+), and
  * Ki67 ≤20% by IHC staining;
* surgically treated with BCS with or without sentinel node biopsy (SNB);
* no clinical evidence of distant metastases. Imaging work up is not mandatory to enter the trial. If there are signs/symptoms suggesting the presence of local relapse or distant metastasis, an appropriate work up should be performed according to the treating physician standard practice. A patient with confirmed local relapse or distant metastasis will no longer be eligible for the trial;
* postoperative final surgical margins negative (no ink on tumor);
* baseline HRQoL questionnaires completion;
* adjuvant bisphosphonates and denosumab are allowed;
* before patient registration/randomization, written informed consent must be given.

Exclusion Criteria:

* Preoperative systemic treatments (i. e., chemotherapy, endocrine therapy);
* current treatment with any hormonal agents such as tamoxifen, raloxifene or other selective estrogen receptor modulators (SERMs), either for osteoporosis or BC prevention (patients are eligible if these medications are discontinued prior to randomization);
* prior breast or thoracic RT;
* known disorders associated with a higher risk for complications following RT such as collagen vascular disease, dermatomyositis, systemic lupus erythematosis or scleroderma;
* prior diagnosis, detection, or treatment of any other invasive cancer (except basal or squamous cell carcinoma of the skin that has been definitely treated);
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; these conditions should be discussed with the patient before registration;
* patients must not be considered a poor medical risk due to serious, uncontrolled medical disorder, non-malignant systemic disease, or active uncontrolled infection. Examples include but are not limited to uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction or uncontrolled major seizure disorder.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 926 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcome measures (PROM) HRQoL as assessed by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 | Change from baseline at 24 months
  EORTC Quality of Life Questionnaire (QLQ) C30.The QLQ-C30 is a cancer HRQoL questionnaire using PROMs for individual patient management. It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Subjects respond on a four-point scale from "not at all" to "very much" for most items. Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function and higher levels of symptom burden.
Time to ipsilateral breast tumor recurrence (IBTR) | 60 months
  Time to ipsilateral breast tumor recurrence (IBTR)

SECONDARY OUTCOMES:
Patient reported outcome measures (PROM) HRQoL as assessed by EORTC Quality of Life Questionnaire (QLQ) BR45 Breast module | Change from baseline at 24 months
  EORTC QLQ BR45 module. The EORTC QLQ BR45 is a breast-specific module that comprises of 45 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss. All scores are linearly transformed to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score. A high QoL is represented by a high score for global health status or QoL. More severe symptoms or problems are represented by high symptom scores or items.
Patient reported outcome measures (PROM) HRQoL as assessed by EORTC Quality of Life Questionnaire (QLQ) ELD14 Elderly module | Change from baseline at 24 months
  EORTC QLQ ELD14 questionnaire. The QLQ ELD14 is a validated HRQoL questionnaire for cancer patients aged ⩾70 years. All scores are linearly transformed to a 0 to 100 scale.
  Five scales: mobility, family support, worries about the future, maintaining autonomy and purpose, and burden of illness. High scores indicate poor mobility, good family support, much worry about the future, good maintenance of autonomy and purpose, and high burden of illness.
Time to locoregional recurrence (LRR) | 24 months
  Time to locoregional recurrence (LRR)
Time to contralateral breast cancer (CBC) | 24 months
  Time to contralateral breast cancer (CBC)
Time to distant metastases (DM) | 24 months
  Time to distant metastases (DM)
Breast cancer specific survival (BCSS) | 24 months
  Rate of death related to breast cancer
Overall survival (OS) | 24 months
  Rate of death related to all causes
Adverse events (AE) | 24 months
  Number of participants with reported AE. The Common Terminology Criteria for Adverse Events (CTCAE) is a descriptive terminology which can be utilized for AE reporting. A grading (severity) scale is provided for each AE term. Grade refers to the severity of the AE. The CTCAE displays Grades 1 (mild) through 5 (death related to AE) with unique clinical descriptions of severity for each AE.
Cosmesis evaluation | 24 months
  Rate of cosmesis assessment grade. The Harvard Breast Cosmesis Scale is a 4-point breast cosmesis grading scale (1. Excellent - 2. Good - 3. Fair - 4. Poor).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, MD,Prof, Study Chair — University of Florence, Florence, Italy; Philip M Poortmans, MD,PhD,Prof, Study Chair — Iridium Kankernetwerk - University of Antwerp; Wilrijk-Antwerp, Belgium; Icro Meattini, MD,Prof, Principal Investigator — University of Florence, Florence, Italy
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi, Florence University, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meattini I, Poortmans PMP, Marrazzo L, Desideri I, Brain E, Hamaker M, Lambertini M, Miccinesi G, Russell N, Saieva C, Strnad V, Visani L, Kaidar-Person O, Livi L. Exclusive endocrine therapy or partial breast irradiation for women aged >/=70 years with luminal A-like early stage breast cancer (NCT04134598 - EUROPA): Proof of concept of a randomized controlled trial comparing health related quality of life by patient reported outcome measures. J Geriatr Oncol. 2021 Mar;12(2):182-189. doi: 10.1016/j.jgo.2020.07.013. Epub 2020 Jul 29. PMID 32739355
- [Background] Meattini I, De Santis MC, Visani L, Scorsetti M, Fozza A, Meduri B, De Rose F, Bonzano E, Prisco A, Masiello V, La Rocca E, Spoto R, Becherini C, Blandino G, Moscetti L, Colciago RR, Audisio RA, Brain E, Caini S, Hamaker M, Kaidar-Person O, Lambertini M, Marrazzo L, Saieva C, Spanic T, Strnad V, Wheelwright S, Poortmans PMP, Livi L; EUROPA Trial Investigators. Single-modality endocrine therapy versus radiotherapy after breast-conserving surgery in women aged 70 years and older with luminal A-like early breast cancer (EUROPA): a preplanned interim analysis of a phase 3, non-inferiority, randomised trial. Lancet Oncol. 2025 Jan;26(1):37-50. doi: 10.1016/S1470-2045(24)00661-2. Epub 2024 Dec 12. PMID 39675376
- [Derived] Ho AY, Bellon JR. Overcoming Resistance - Omission of Radiotherapy for Low-Risk Breast Cancer. N Engl J Med. 2023 Feb 16;388(7):652-653. doi: 10.1056/NEJMe2216133. No abstract available. PMID 36791166